CLINICAL TRIAL: NCT02869061
Title: Effectiveness and Safety of Local Endoscopically-assisted Administration of Autologous Adipose-derived Regenerative Cells for Reduction of Risk of Postoperative Bladder Neck Contracture in Male Patients
Brief Title: Effectiveness and Safety of Adipose-derived Regenerative Cells for Reduction of Risk of Bladder Neck Contracture
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RU-CCH-01-02-15
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Bladder Neck Obstruction; Bladder Outlet Obstruction; Benign Prostatic Hyperplasia; Urinary Bladder Neck Obstruction
Keywords: Bladder neck obstruction; Bladder outlet obstruction; Benign prostatic hyperplasia; Urinary bladder neck obstruction; Bladder neck contracture; Bladder neck stricture; Bladder neck stenosis; Transurethral resection of the prostate; Prostatectomy; Stromal vascular fraction (SVF); Adipose-derived regenerative cells (ADRC); Adipose tissue; Stem cells
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Prostatic Hyperplasia | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADRC injection (Experimental): Subjects will be undergone liposuction under local anesthesia. Adipose-derived regenerative cells (ADRC) will be isolated from lipoaspirate by enzymatic digestion. Transurethral bladder neck resection followed by the injection of ADRC suspension will be performed. This is a single arm study with no control. All patients receive cell therapy.
  Interventions: Procedure: Liposuction; Procedure: Transurethral bladder neck resection.; Biological: ADRC; Other: ADRC isolation

INTERVENTIONS:
Procedure: Liposuction
Procedure: Transurethral bladder neck resection.
Biological: ADRC — Injection of ADRC suspension will be performed endoscopically into the bladder neck close to the site of resection.
  Other Names: Adipose-derived regenerative cells
Other: ADRC isolation — ADRC will be isolated according to patent pending technology based on enzymatic digestion, washing and concentration of cell pellet in up to 9.5 ml of normal saline.

SUMMARY:
Autologous adipose-derived regenerative cells (ADRC) will be extracted from lipoaspirate by enzymatic digestion from a portion of the fat harvested from the patient's front abdominal wall. Transurethral bladder neck resection followed by the injection of ADRCs suspension will be performed. This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Fat tissue obtainment:

Subjects will undergo liposuction under local anesthesia. In this procedure, Ringer's solution with the anesthetic lidocaine and vasoconstrictor adrenaline infused into the adipose compartment to minimize blood loss and contamination of the tissue by peripheral blood cells. 15 minutes later a hollow blunt-tipped 3 mm cannula introduced into the subcutaneous space through small (0.5 cm) incision. The cannula attached to syringe and under gentle suction moved through the adipose compartment, mechanically disrupting the fat tissue. Aspirate volume - approximately 150-200 cc. Procedure time - 30 minutes.

ADRC isolation:

Harvested adipose tissue will be processed according to patent pending technology based on enzymatic digestion, washing and concentration of cell pellet in 9.5 ml of normal saline.Obtained ADRC divided into 2 portions. First portion (0.5 mL) used for counting, viability and sterility assessment. The second portion (9 ml) placed into sterile syringe for injection.

Surgery:

Transurethral endoscopic loop resection of bladder neck will be performed.

Autologous ADRC administration:

Injection of ADRC suspension will be performed immediately after bladder neck resection. 9 to 18 injections (0.5 to 1.0 mL each) will be injected with endoscopic needle into the bladder neck close to the site of resection. All injections will be performed during single procedure.

ELIGIBILITY:
Inclusion Criteria:

* Bladder neck contracture after transurethral prostate resection.
* Obstructive pattern of urine flow rate with maximum flow rate below 15 mL/s
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Contraindications for spinal, epidural or inhalation anesthesia
* Urethral strictures
* Genitourinary inflammatory diseases
* Prostate-specific antigen (PSA) level above 4 ng/mL
* Contraindications for local anesthesia or history of allergy for local anesthetics
* Systemic glucocorticoid and/or immunosuppressant therapy
* Any condition that might limit compliance (dementia, mental disorders, narcotic drug or alcohol abuse etc.)
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy
* Clinically significant abnormalities in results of laboratory tests
* Patient received anticoagulants at least 12 hours prior the liposuction
* Medical history of heterotopic ossifications
* Patients prescribed for glycoprotein inhibitors treatment

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Chronic kidney disease IV- V stages (creatinine clearance < 30 mL/min estimated by Cockcroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | 4 weeks after injection of ADRC suspension
  Frequency, type and severity of serious adverse events (SAE)
Serious adverse reactions | Time Frame: 4 weeks after injection of ADRC suspension
  Frequency, type and severity of serious adverse reactions (SAR)

SECONDARY OUTCOMES:
Changes of the volume of residual urine | Follow up to completion (48 weeks after intervention)
  Influence of the procedure on the volume of residual urine assessed by ultrasonography
Urodynamic changes - 1 | Follow up to completion (48 weeks after intervention)
  Influence of the intervention on urinary flow rate: maximum flow rate
Urodynamic changes - 2 | Follow up to completion (48 weeks after intervention)
  Influence of the intervention on urinary flow rate: average flow rate
Urodynamic changes - 3 | Follow up to completion (48 weeks after intervention)
  Influence of the intervention on urinary flow rate: total volume voided
Urodynamic changes - 4 | Follow up to completion (48 weeks after intervention)
  Influence of the intervention on urinary flow rate: maximum flow time
Quality of life monitoring - 1 | Follow up to completion (48 weeks after intervention)
  Quality of life estimated by validated questionnaire: the Short Form (SF-36).
Quality of life monitoring - 2 | Follow up to completion (48 weeks after intervention)
  Quality of life estimated by validated questionnaire: International Prostatic Symptom Score (IPSS).
Bladder neck restenosis control | Follow up to completion (48 weeks after intervention)
  Revision of bladder neck structure by retrograde urethrography

CONTACTS AND LOCATIONS:
Overall Officials: Denis V Butnaru, MD, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University; Andrey A Pulin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Andrey Z Vinarov, MD, PhD, Prof, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (2):
- Russia (2):
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation, Moscow

IPD SHARING:
Plan to Share IPD: Undecided